CLINICAL TRIAL: NCT01054287
Title: Falls Prevention Program in Acute Care Hospital
Brief Title: Falls Prevention in Acute Care Hospital
Acronym: PRECEPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Other Study IDs: SQO150
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Falls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Falls prevention (Experimental)
  Interventions: Other: Multifactorial falls prevention program
- Usual care (Placebo Comparator)
  Interventions: Other: No falls prevention intervention

INTERVENTIONS:
Other: Multifactorial falls prevention program
  Arms: Falls prevention
Other: No falls prevention intervention
  Arms: Usual care

SUMMARY:
The aim of this study is to evaluate the effect of a multifactorial falls prevention program in an acute internal medicine ward.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to internal medicine ward

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
falls rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Service of internal medicine, CHUV, Lausanne, Canton of Vaud, Switzerland